CLINICAL TRIAL: NCT06757192
Title: Initiating Colorectal Cancer Screening in Unscreened Individuals 45 to 54
Brief Title: CRC Screening in Unscreened Individuals 45-54
Status: Recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: American College of Gastroenterology (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Adjoa Anyane-Yeboa, M.D., Principal Investigator, Massachusetts General Hospital
Other Study IDs: 24-219
Record Dates: First submitted 2024-12-05; First posted 2025-01-03 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Cancer Screening
Keywords: colorectal cancer screening

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients and staff from one community health center named Codman Square Health Center.: This project builds on an existing partnership with Codman Square Health Center (CSHC). CSCHC is located in the Dorchester neighborhood of Boston which has among the highest mortality rates from colorectal cancer in the city. Codman Square Health Center serves a patient population that is 86% Black and 87% income at or below the federal poverty limit, thus requiring an equity-driven approach. Patients recruited will be aged 45-54 and staff will be over aged 18 who work at CSHC and that are involved in CRC screening. There will be no clinical intervention as this is an implementation study to identify system-level determinants of colorectal cancer screening.

SUMMARY:
The goal of this observational study is to understand the barriers and facilitators to completing colorectal cancer screening from the patient and community health center staff perspective. The main question it aims to answer is to identify system-level determinants of colorectal cancer screening in individuals aged 45 to 54. Participants will be asked to partake in one-time interviews either online or in-person and community health center staff will also be asked to take an online survey.

DETAILED DESCRIPTION:
AIM 1: Identify system-level determinants of CRC screening in individuals age 45 to 54 using mixed methods.

A. Overview: The objective of this aim is to identify systems-level determinants of CRC screening in unscreened individuals age 45 to 54 at CSHC using the CFIR framework. We will work with Dr. Rachel Hindin, our clinical champion, to: (1) conduct a validated organizational survey with staff and providers and connect to patient-level EHR data to quantitatively assess systems-level determinants of screening; (2) conduct in-depth interviews with patient-facing CHC staff and providers; and (3) conduct in-depth interviews with patients.

B. Approach: B.1. Organizational Survey: Participants and recruitment: The organizational survey will be conducted at CSHC and 9 other CHCs, which will allow us to gather generalizable information about systems-level determinants of screening (n(CHCs) = 10; n(survey participants) = 50; n=5 staff and providers directly involved in CRC screening per CHC). Eligible staff at CHCs will be identified by our staff contact at each CHC.

Procedures: We will use a validated survey previously developed by ISCCCE, to collect data on systems-level factors that contribute to CRC screening. The survey collects data on CFIR inner setting constructs at the CHC including human resources practices, learning climate, available resources, patient needs and resources, linguistic services, implementation demands, and leadership engagement. Survey data will be collected via RedCap. Electronic informed consent will be obtained prior to each survey. Written or phone surveys (written or verbal consent) will be offered to those unable to provide electronic responses. We will connect survey data with patient DRVS data and fit models to quantitatively determine independent systems-level determinants of CRC screening. We will collect data across 10 ISCCCE partner sites which will also allow us to identify sites within the Mass League with similar contexts for testing in my future R01 and to maximize generalizability.

Data Analysis: Characteristics will be measured using a 5-point Likert scale with a "1" rating meaning strongly disagree and "5" rating meaning "strongly agree." Scores across responses will be collected as mean and standard deviations, and an aggregate score will be created by averaging survey responses pertaining to each characteristic. Generalized linear mixed effect models will be used to examine the outcome of CRC screening (yes/no) as function of patient demographics (first level) and inner setting survey construct scores (second level). Findings from the organizational survey will be used to adapt staff and patient interview guides to allow us to dive deeper into findings from the survey. Prior to the start of analysis, I will complete coursework in multilevel modeling under the guidance of Dr. Chan.

In-depth interviews: Participants and recruitment: We will conduct in-depth interviews with a sample of providers and staff (n=10, 5 who took organizational survey) directly involved in CRC screening practices in patient-facing roles and 10 interviews with patients per age strata (n=10 45-49; n= 10 age 50-54). We will ensure an equal sample of screened and unscreened patients amongst each stratum. Patients aged 45 to 54 years who have been seen in the primary care clinic within the last 36 months and are average-risk for CRC (e.g. no family or personal history of CRC, no high-risk cancer syndromes such as Lynch Syndrome, no history of inflammatory bowel disease) will be recruited for in-depth interviews. We will ensure race/ethnicity and sex distribution (male/female) proportionate to the clinic demographics. We expect that 20 interviews with patients and 10 interviews with staff will lead to thematic saturation, but will extend if needed. Eligible staff will be identified by Dr. Hindin; eligible patients will be identified by their providers and contacted by the study team.

Procedures: Informed consent will be obtained prior to each interview (written for in-person and verbal for video interviews). I will conduct interviews, with Dr. Park observing and providing feedback. I will complete interviewer training from the Qualitative and Mixed Methods Research Unit at MGH and pilot the interview guide with the research team and a separate sample of representative patients (using recruitment and consent procedures as above) prior to conducting interviews. Each interview will be audio-recorded with participants' permission, and sessions will be conducted in-person or via video based on participant preference.

Content of CFIR inner setting questions will be informed by organizational survey findings. Guided by CFIR 2.0, qualitative domains for patient interviews will include 1) The Innovation (e.g., knowledge/perceptions about CRC screening); 2) Outer Setting (e.g., structural barriers to screening); 3) Inner Setting (e.g., provider recommendation regarding CRC screening); 4) Characteristics of Individuals (e.g. knowledge/attitudes about preventive health behaviors). The CFIR qualitative interview domains for staff interviews will include 1) The Innovation (e.g., knowledge/perceptions about CRC screening); 2) Outer Setting (e.g., structural barriers to screening, public awareness about screening); 3) Inner Setting (e.g., leadership and staff buy-in, resources, patient needs); 4) Characteristics of Individuals (e.g. linguistic representation, staff turnover); 5) Implementation Process (implementation stress/demands).

Data Analysis: I will oversee all data collection and analysis. Interviews will be recorded and transcribed using an institutionally-approved software and analyzed using NVivo. Analyses will include inductive (thematic analyses of barriers and facilitators) and deductive strategies (structural coding). We will apply the 5 stages of Framework analyses (Familiarization, Identifying Themes, Indexing, Charting, and Interpreting)48 to conduct content analyses, which will be done by me and a research coordinator with oversight from Dr. Park. We will analyze along CFIR domains. Discrepancies will be resolved with Dr. Park through discussion and comparison of raw data. Coding will continue until a high level of reliability (Kappa=>0.80) is established. Qualitative findings will be compared by age-specific strata for patients, and patients vs staff. Prior to interviews, I will complete coursework in qualitative analysis.

Expected Outcomes: The identification of system-level determinants of CRC screening. Potential Problems and Alternative Strategies: A potential problem may be difficulty recruiting patients for interviews. Recruitment will be done with the help of Dr. Hindin, our clinical champion who has prior success in recruiting individuals for qualitative data collection

AIM 2: Identify equity-driven implementation strategies to initiate CRC screening.

A. Overview: Aim 2 will match systems-level determinants (from Aim 1) to potential implementation strategies.

B. Approach: B.1. Workflow mapping: After determinant themes are identified, we will meet with Dr. Hindin and her team for workflow mapping. Workflow maps detail every step in the CRC screening process and identify where new strategies will fit in the workflow.

B.2. Implementation Strategy Development: Implementation road maps will be used to develop implementation strategies49. The roadmaps are causal loop diagrams that are used to develop a single implementation strategy matched to a specific determinant. We will first rank determinants (high/medium/low). We will then develop implementation roadmaps focused on high-ranking determinants, identify a plausible strategy to address the identified determinant, report proximal and distal outcomes, and identify moderators that could impact the likelihood that each step in the causal pathway will take place. Multiple roadmaps will be developed based on identified determinants and we will develop a list of potential implementation strategies based on ranking, CHC needs, and preferences. Expected Outcomes: The identification of systems-level implementation strategies matched to barriers specific to CHC needs and resources.

D. Potential Problems & Alternative Strategies: Strategies may not fit into existing workflows or may add burden. In this case, we will determine if new workflows can be created, or if a different strategy is needed.

E. Timeline and Deliverables: Aim 2 activities will occur in Year 3 and will result in 3 manuscripts.

AIM 3: To determine the acceptability and feasibility of implementation strategies for CRC screening by conducting a pilot trial and using mixed methods.

A. Overview: Aim 3 will test systems-level implementation strategies (identified in Aim 2) matched to systems-level determinants of CRC screening (Aim 1) at CSHC and evaluate outcomes using mixed methods. Approach: B.1. Population: Individuals aged 45 to 54 who are newly eligible or have never been screened for CRC will be identified using the DRVS platform. DRVS allows for population management views of individuals who are due for cancer screening. There are 4,384 patients at CSHC age 45 to 54 and 1,599 who are unscreened and eligible for inclusion.

B.2.Study Design: We will test the 2 highest ranking barrier-strategy combinations (identified in Aims 1 and 2). We will test each barrier-strategy combination separately for a total of 12 months. The most feasible and acceptable strategies will continue to be used and sustainability will be measured 6 months after completion of the last cycle. Data Collection: C.1.Quantitative data: Data will be collected via Redcap survey and electronic health record.

C.2.Qualitative data: One-on-one semi-structured interviews will be conducted with staff who filled out surveys (n = 15) to further explore the acceptability and feasibility, reach, effectiveness, successes, and challenges faced. Data on maintenance of program components will be collected at 6 months post-pilot. Interviews will be 1 hour in duration and conducted in person or over Zoom video conference. Interview guides will be structured following RE-AIM and adapted to explore survey findings in greater depth using an explanatory sequential mixed methods design. Consent for surveys and in-person or video interviews will be the same as in Aim 1. Data Analysis: D.1.Quantitative data: For our primary outcome, participants will be asked to rate the acceptability and feasibility of implementation strategies using a previously validated instrument50, which we have previously used with CHC staff. This tool has demonstrated good internal consistency reliability (0.85 for acceptability and 0.89 for feasibility) and similarly good test-retest reliability (correlations: acceptability- 0.80; feasibility - 0.88) and validity in a known groups analysis50. There is no established acceptability and feasibility benchmark for these measures. Quantitative data will provide a numeric summary of acceptability and feasibility which will inform the development of interview guides for qualitative data collection. For secondary outcomes, descriptive statistics (relative frequencies, means, variability) will be used to evaluate reach (the number of patients offered CRC screening measured by calculating the number of patients with a FIT order or colonoscopy referral during the pilot testing period), effectiveness (time to CRC screening measured by assessing the difference in the date CRC screening was completed compared to the start date of pilot testing and number screened for CRC pre and post intervention), and maintenance (percentage of program components maintained). We will use generalized linear models to estimate the level of effectiveness, reach, and maintenance across clinical characteristics and sociodemographics with a particular focus on characteristics around equity. Given the limited time frame for testing of each strategy and drawing on the literature51-54, we will use a 10% increase in overall screening, at this predominantly Black CHC, as our target indicator of advancing equity. We will also explore differences in equity outcomes among subgroups, recognizing that our power is limited.

D.2.Qualitative data: We will follow the same framework analysis as AIM 1, using RE-AIM domains.

Consistent with the purpose and intent of a pilot study as described in detail by Leon and Kramer and colleagues55,56, our study will evaluate feasibility, acceptability, and potential effectiveness but will not be powered to test statistical significance or to formally test a hypothesis, which will be the intent of my future R01. E. Potential Problems & Alternative Strategies: A potential challenge may be getting staff to fill out surveys with outcome assessments in a timely manner after each cycle. If this occurs, we will send reminders in emails, at staff meetings, offer verbal surveys, and consider small incentives (e.g. $35 gift cards) for survey completion.

ELIGIBILITY:
PATIENTS

Inclusion Criteria:

* Individuals aged 45-54
* Individuals who are patients at the health center
* Individuals that are willing and able to give verbal/written consent

Exclusion Criteria:

* Individuals with a personal history of CRC
* Individuals with a family history of CRC
* Individuals with a history of inflammatory bowel disease or high-risk cancer syndrome

STAFF

Inclusion Criteria:

* Individuals ages 18+
* Individuals working at the health center
* Individuals that are involved in CRC screening processes at CSHC
* Individuals that are willing and able to give verbal/written consent

Ages: 45 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Survey participants will involve staff members and providers (ages 18+) involved with CRC screening processes. Patients will be health center patients.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2029-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Measurement of acceptability and feasibility of implementation strategies | From planning to testing and evaluation and assessment of outcomes will be a total of 12 months
  For our primary outcome, participants will be asked to rate the acceptability and feasibility of implementation strategies using a previously validated instrument, which the investigator previously used with CHC staff. This tool has demonstrated good internal consistency reliability (0.85 for acceptability and 0.89 for feasibility) and similarly good test-retest reliability (correlations: acceptability- 0.80; feasibility - 0.88) and validity in a known groups analysis. There are no cut off numbers for acceptability and feasibility as these are just means but higher scores reflect higher acceptability. However, our surveys will allow us to better understand our survey findings. Quantitative survey interviews will be collected after first and second cycle of testing. The surveys and interviews will be measured together as this is a mixed methods study.

SECONDARY OUTCOMES:
Measurement of reach, effectiveness, and maintenance of implementation strategies | From planning to testing and evaluation and assessment of outcomes will be a total of 12 months
  For secondary outcomes, descriptive statistics (relative frequencies, means, variability) will be used to evaluate reach (the number of patients offered CRC screening measured by calculating the number of patients with a FIT order or colonoscopy referral during the pilot testing period), effectiveness (time to CRC screening measured by assessing the difference in the date CRC screening was completed compared to the start date of pilot testing and number screened for CRC pre and post intervention), and maintenance (percentage of program components maintained). The investigator will use generalized linear models to estimate the level of effectiveness, reach, and maintenance across clinical characteristics and sociodemographics with a particular focus on characteristics around equity. This is a mixed methods study where interviews and descriptive statistics will be measured together as mixed methods study.

CONTACTS AND LOCATIONS:
Overall Officials: Adjoa Anyane-Yeboa, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Codman Square Health Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided